CLINICAL TRIAL: NCT02806492
Title: Blood Pressure or Cardiac Output - the Influence on Cerebral Perfusion During Cardiopulmonary Bypass
Brief Title: Parameters of Cerebral Perfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Dr. B. van Zaane, MD PhD, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL48417.041.14
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Cerebral Perfusion; Cerebral Oxygenation; Cardiopulmonary Bypass
MeSH Terms: interventions — Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient for cardiac surgery (Experimental): All patient undergo the 5 different intervention in a randomised matter.
  Interventions: Other: 50-100ug phenylephrine before CPB; Other: 50-100ug phenylephrine during CPB; Other: decreasing CPB flow; Other: Decreasing CPB flow AND 50-100ug phenylephrine; Other: Increasing CPB flow

INTERVENTIONS:
Other: 50-100ug phenylephrine before CPB — In this intervention we will administer 50-100 μg phenylephrine to the patient before CPB is started. This intervention will take place when the patient shows hypotension (MAP <60mmHg, according to protocol22). Because of the increase in PVR there will be a baroreceptor-reflex-mediated decrease in CO. On-line, we will quantify the percentage decrease in systemic blood flow (i.e. CO) by using the Modelflow algoritm incorporated in a non-invasive beat-to-beat finger blood pressure monitor. This will allow us to obtain a reference for the decrease in CO to use in the next interventions. Our hypothesis is that CO will decrease because of the baroreceptor-reflex. During this intervention NIRS and TCD MCA will be recorded.
Other: 50-100ug phenylephrine during CPB — In this intervention we will induce only 1 component of the changes at intervention (1), being the increase in MAP of approximately 20 mmHg by administrating 50-100 μg phenylephrine. The CPB enables us to maintain a constant CO and thus eliminating the baroreceptor-reflex. During this intervention NIRS and TCD MCA will be recorded.
Other: decreasing CPB flow — With this intervention we will only create a change in CO, which enables us to eliminate the effect of blood pressure. We will modify CPB flow to achieve the CO decrease (in %) measured at intervention (1) meaning: pre-CPB after the bolus of 50-100 μg phenylephrine. In the case of unexpected increase (in %) of CO measured at intervention (1), we will still decrease CPB flow so we will be able to analyse decrease as well as increase in CPB flow. During this intervention NIRS and TCD MCA will be recorded.
Other: Decreasing CPB flow AND 50-100ug phenylephrine — In this intervention we will simulate the 'normal' physiological state when administering phenylephrine. We will modify CPB flow to achieve the percentage change CO as observed during intervention (1) as well as administrate 50-100 μg phenylephrine. We expect to see similar outcomes as in intervention (1). During this intervention NIRS and TCD MCA will be recorded.
Other: Increasing CPB flow — In this last intervention we will create an increase in MAP without using phenylephrine but only by increasing CO. This enables us to eliminate a possible direct α1-adrenergic effect on the cerebral vasculature. MAP will be raised approximately 20 mmHg by increasing CPB flow 20%. During this intervention NIRS and TCD MCA will be recorded.

SUMMARY:
The purpose of this study is to determine whether cerebral blood flow and cerebral tissue oxygenation is most dependent on cardiac output or on mean arterial pressure in patients undergoing cardiac surgery with the use of cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiopulmonary bypass for CABG a
* having an appropriate temporal bone window for reliable TCD monitoring
* needing pharmacological intervention because of hypotension before going on CPB.

Exclusion Criteria:

* requiring hypothermia during surgery
* requiring emergency surgery
* contraindication for phenylephrine,
* having known brain pathology (e.g. Cerebral Vascular Accident (CVA) or increased intracranial pressure
* having a history of severe carotid artery stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
regional cerebral oxygen saturation | During surgery
mean velocity of blood flow of the middle cerebral artery | During surgery

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands